CLINICAL TRIAL: NCT04002622
Title: A Phase II, Multicenter, Open, Single-arm Study of TQB2450 Injection (PD-L1 Antibody) in Subjects With Relapsed or Refractory Primary Mediastinal B-cell Lymphoma (rrPMBCL)
Brief Title: Study of TQB2450 Injection in Subjects With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The population of target indication is small and screening is difficult.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-02
Record Dates: First submitted 2019-06-27; First posted 2019-06-28 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Relapsed or Refractory Primary Mediastinal B-cell Lymphoma (rrPMBCL)
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450 (Experimental): TQB2450 1200 milligrams (mg) administered intravenously (IV) on Day 1 of each 21-day cycle.
  Interventions: Drug: TQB2450

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

SUMMARY:
TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed relapsed or refractory primary mediastinal large B-cell lymphoma.

  2. 18 and 75 years; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy > 3 months.

  3. At least one measurable lesion. 4. Left ventricular ejection fraction (LVEF) measured by the cardiac echocardiography ≥ 50%.

  5. Screening laboratory values must meet the following criteria:hemoglobin ≥ 80 g/L; neutrophils ≥ 1.5*10^9/L; platelets ≥ 100 x 10^9/ L.

  6. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Abm or its components.

  2. Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody ,or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.

  3. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks.

  4. Has received emergency cytoreductive surgery to control tumors. 5. Has received allogeneic hematopoietic stem cell transplantation within the last 5 years.

  6. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  7. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include basal cell skin cancer, squamous cell carcinoma of skin, melanoma skin and cancer carcinoma in situ of the cervix.

  8. Has definite central nervous system (CNS) infiltration of lymphoma, including brain parenchyma, meningeal invasion or spinal cord compression.

  9. Has any active autoimmune disease or a history of autoimmune disease. 10. Has serious or uncontrolled diseases such as history of chronic heart failure.

  11. Has any active autoimmune disease or a history of autoimmune disease. 12. Has received blood transfusion, erythropoietin granulocyte colony stimulating factor(G -CSF)，or Granulocyte macrophage colony stimulating factor(GM-CSF) within 4 weeks before the first dose.

  13. Has vaccinated with vaccines or attenuated vaccines within 4 weeks before the first dose.

  14. Has received surgery, or unhealed wounds within 4 weeks before the first dose.

  15. Has Hepatic, renal, blood coagulation dysfunction. 16. Has interstitial lung disease or non-infectious pneumonia and present residual lesions.

  17. Has received systemic treatment for active infection before the first dose.

  18. Has active or latent tuberculosis. 19. Hepatitis B virus surface antigen (HBsAg) positive, and hepatitis B virus DNA copy number > upper limit of normal.

  20. Human immunodeficiency virus antibody positive , hepatitis C antibody (HCV-Ab) and hepatitis C virus DNA copy number > upper limit of normal.

  21. Breastfeeding or pregnant women. 22. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 96 weeks
  Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Disease Control Rate (DCR) | up to 24 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Time to Response (TTR) | up to 24 months
  TTR defined as time from the first dose to the first assessment of PR or CR.
Overall Survival (OS) | up to 24 months
  OS defined as the time from randomization to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fifth Medical Center of the Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijin, Beijing Municipality
  - Peking Hospital, Beijin, Beijing Municipality
  - Union Medical College Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan People's Hospital, Zhengzhou, Henan
  - Hunan Canser Hospital, Changsha, Hunan
  - First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Tongji Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tumor Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Tumor Hospital, Hangzhou, Zhejiang